CLINICAL TRIAL: NCT04323566
Title: A Randomized, Double-blinded, Placebo-controlled Study of Rituximab in Patients with Psychosis And/or Obsessive Compulsive Disorder, with an Indication of Immune System Involvement
Brief Title: Rituximab Treatment for Psychosis And/or Obsessive Compulsive Disorder with Probable Immune System Involvement
Acronym: Ra-P-OCD
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Janet Cunningham, MD Associate Professor Janet Cunningham, Uppsala University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ra-P-OCD 1.2, 2020-02-04; 2024-518391-31-00 (EU CTIS Number); 2019-000256-33 (EudraCT Number)
Record Dates: First submitted 2020-03-10; First posted 2020-03-26 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Obsessive-Compulsive Disorder; Obsessive-Compulsive Behavior; Schizophrenia; Delusional Disorder; Brief Psychotic Disorder; Schizo Affective Disorder; Other Psychoses; Unspecified Psychosis
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Compulsive Behavior; Schizophrenia; Schizophrenia, Paranoid; Psychotic Disorders; Mental Disorders | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: This is a placebo-controlled, interventional study of parallel groups with 40 participants, randomized to either treatment-first with 500 mg Rituximab i.v. at 0 (infusion 1) and at 4 months (infusion 2), or placebo-first, with NaCl-infusions at 0 and at 4 months. Main evaluation takes place at eight months. The study arms are then crossed over, i.e. those with treatment-first receive placebo at 8 (infusion 3) and 12 months (infusion 4), and those with placebo-first receive Rituximab at these time points. Final evaluation takes place at 16 months. Before each infusion, all patients are pre-treated with Solu-Medrol i.v., Paracetamol p.o. and Cetirizin p.o. Patients are monitored with psychiatric rating scales and blood samples at baseline (-1 month) and every four months. The evaluations at baseline, eight and 16 months also encompass collection of CSF (lumbar puncture), psychologic testing and extended blood samples.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The nurse(s) administering Rituximab or placebo (NaCl) infusions will be prevented from having insight into which of the infusions she/he is administering.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment-first arm (Experimental): Participants receive i.v. infusions with 500 mg Rituximab at 0 and 4 months, followed by placebo infusions (NaCl) at 8 and at 12 months, Pre-treatment prior to all four infusions consists of injection Solu-Medrol 125 mg i.v., tablet Paracetamol 1000 mg p.o. and tablet Cetirizin 10 mg p.o.
  Interventions: Drug: Rituximab
- Placebo-first arm (Experimental): Participants receive placebo (NaCl) i.v. infusions at 0 and 4 months, followed by 500-mg-Rituximab infusions at 8 and 12 months. Pre-treatment prior to all four infusions consists of injection Solu-Medrol 125 mg i.v., tablet Paracetamol 1000 mg p.o. and tablet Cetirizin 10 mg p.o.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab 500 mg, dissolved in 250 ml NaCl in an infusion bag, covered with non-see-through plastic
  * administered iv over a course of max 180 minutes
  * at 0 and 4 months (treatment-first arme) OR at 8 and 12 months (placebo-first arm)

SUMMARY:
The primary objective for this study is to evaluate whether Rituximab as compared to placebo is a clinically effective treatment for a subgroup of patients suffering from psychosis and/or obsessive-compulsive disorder (OCD) or -behavior (OCB) where there is an indication of immune system involvement.

The secondary objectives of this study are

1. To assess whether Rituximab treatment (with the doses and timing described below) as compared to placebo is associated with amelioration in psychiatric symptomatology
2. To assess whether Rituximab treatment as compared to placebo is associated with improvement in executive functions
3. To assess whether Rituximab treatment as compared to placebo is associated with amelioration in neurological symptoms
4. To evaluate the longevity of psychiatric, neurological and executive improvements associated with Rituximab treatment for up to 16 months after the first infusion (i.e. 12 months after the last infusion)
5. To evaluate whether Rituximab treatment as described is safe for these patients.

The exploratory objectives of this study are

1. To assess changes in blood and cerebrospinal fluid (CSF) markers for immune activity associated with Rituximab treatment compared to placebo
2. To assess statistical associations between biological markers in blood or CSF and clinical response
3. To describe changes in somatic symptoms associated with treatment with Rituximab vs placebo for patients with initial symptoms in the questionnaires
4. To describe changes on MR and EEG associated with treatment with Rituximab vs placebo for patients with initial pathology in these examination
5. To study immune mechanisms coupled with psychiatric symptoms, possibly identifying novel biomarkers with potential for subtyping encephalopathies with immune engagement, using biobank cells, blood and CSF samples collected from the participants.

DETAILED DESCRIPTION:
METHODOLOGY:

This study is planned as a placebo-controlled, interventional study of parallel groups with 40 participants. Patients will be randomized to either treatment-first arm with 500 mg Rituximab i.v. (infusion 1) at 0 and again at 4 months (infusion 2), or placebo-first arm, receiving NaCl-infusion at 0 and at 4 months. Main evaluation will take place at eight months. The study arms are switched after eight months, i.e. patients starting in the treatment-first arm will receive placebo (NaCl) infusions at 8 months (infusion 3) and 12 months (infusion 4), and patients in the placebo-first arm receive 500 mg-Rituximab infusions at these time points. Final evaluation is scheduled at 16 months. Before each infusion, all patients in the Rituximab and control groups are pre-treated with injection Solu-Medrol 125 mg, i.v., tablet Paracetamol 1000 mg, p.o. and tablet Cetirizin 10 mg, orally.

Patients will be monitored with psychiatric rating scales and blood samples at baseline and every four months. In addition, baseline (-1 months), main (8 months) and final evaluation (16 months) will encompass collection of CSF (lumbar puncture), psychologic testing and extended blood samples. Patient, nurse administering treatment and symptom evaluators are blinded to group randomization.

INVESTIGATIONAL PRODUCT, DOSAGE AND MODE OF ADMINISTRATION:

* Treatment: Rituximab (Roche), 500 mg, dissolved in 250 ml NaCl 9 mg/ml, administered intravenously twice with 4 months interval.
* Placebo: 250 ml NaCl 9 mg/ml, administered intravenously twice with 4 months interval.

Duration of treatment:

Patients are observed over the course of 16 months. Main evaluation is conducted after 8 months. Participants are randomized to either treatment-first (Rituximab infusion at 0 months and 4 months) or placebo-first (Rituximab infusion at 8 months and 12 months).

SITE MONITORING AND SOURCE DATA VERIFICATION

The Investigator(s)/institution(s) will permit study-related monitoring, audits, review and regulatory inspection(s), providing access to source data/hospital records. Sponsor verifies that each patient has consented in writing to direct access to the original source data/hospital records by the use of written patient information and signed Informed Consent.

In accordance with the principles of Good Clinical Practice (GCP), monitoring of the study will be arranged by the Sponsor. During the study, the Monitor will have regular contacts with the study site(s), including visits to ensure that the study is conducted and documented properly in compliance with the protocol, GCP and applicable regulatory requirements.

Prior to the start of the study, the monitor will review the protocol and CRFs with the investigator and his/her staff. The investigator will be visited by the monitor, who will check study procedures, including safety assessments, study medication handling, and data recording.

To assure the accuracy and completeness of the data recorded in the trial, the monitor will compare Case Report Forms (CRFs) with medical records and other relevant documentation during the on-site monitoring visits (source data verification, SDV). The monitor will have direct access to all source data according to International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) GCP. Incorrect or missing entries into the CRFs will be queried and must be corrected. Any discrepancies of data will be documented and explained in the monitoring reports. Study monitoring will not jeopardize patient confidentiality.

The study center may also be subject to inspection by the Swedish Medical Products Agency (MPA). The Investigator and other responsible personnel must be available during the monitoring visits and a possible inspection, and should devote sufficient time to these processes.

DATA COLLECTION AND MANAGEMENT

Data management and handling of data will be conducted according to the study specific Data Management Plan with ICH guidelines and an assigned CRO's standard operating procedures (SOPs). An electronic CRF (eCRF) system will be used to capture data from the study. Data entry will be performed by the study site personnel. Validation and data queries will be handled by the CRO's Data Management Team. The data will be subjected to validation according to the CRO's SOPs in order to ensure accuracy in the collected CRF data.The CRF will have an audit trail with appropriate functionality for data capture, tracking and documentation of any queries or changes. Electronic signatures will be used to lock the data and identify the person entering or changing the data.

Before database closure a reconciliation will be performed between the Serious Adverse Events (SAEs) entered in the safety database and the study database. After database closure, the database will be exported as Statistical Analysis System (SAS®) data sets. Any discrepancies and additions from the process defined in the Data Management Plan, will be described in a study specific Data Management Report.

STATISTICAL ANALYSIS:

The trial comprises a fully blinded randomized part, up to and including the 8 month visit, and a follow-up part, with preserved blinding but where it is known that the patient has received Rituximab treatment either in the fully blinded part of the trial or in the follow-up part. The main treatment comparisons will be based on the fully blinded 8 months of the trial, analyzed as a parallel group trial as described below. Data from the follow-up part will be presented descriptively and will be used for explorative modelling of treatment response and duration.

ANALYSIS POPULATION:

The full analysis set (FAS) will consist of all randomized patients that received at least one dose of investigational treatment, and will be used for all analyses unless specified. The number of patients with available data for each outcome analysis will be tabulated. In baseline-adjusted analyses, patients that lack baseline data will be excluded.

DESCRIPTIVE STATISTICS:

Brief Psychiatric Rating Scale (BPRS) score over time, for both parts of the trial, will be described using time series plots of individual data and randomized treatment arm mean values. BPRS and BPRS linear change from baseline at each time point will be described by randomized treatment using dot plots, scatter plots with baseline value on the x-axis, and tables of mean, standard deviation, median, min, max and quartiles.

PRIMARY ANALYSIS:

The primary outcome, BPRS at 8 months, will primarily be analyzed using a linear model with randomized treatment and baseline BPRS as covariates, and presented as the mean difference between the treatment groups with 95% confidence interval (CI) and two-sided p-value. Primarily the analysis will be based on observed cases, which gives unbiased estimation under a mechanism with random missingness conditional on baseline BPRS and treatment arm.

SENSITIVITY ANALYSES:

* To address missing data,

  1. primary analysis with missing 8-month values imputed by the 4-month value when available, and the baseline value otherwise. Under a scenario of no increase in BPRS over time and drop-out mainly due to lack of effect, this analysis would be biased against superiority of the Rituximab treatment.
  2. analyses of a continuum of scenarios based on a model assuming a treatment group dependent missingness propensity estimated from the observed frequencies, and a treatment group dependent difference in baseline-adjusted mean BPRS between observed and missing outcomes. The results will be presented as contour plots of point estimates, lower and upper 95% CI limits, and 2-sided p-values, for each pair of treatment arm specific differences between observed and missing outcomes. The results will indicate what mean deviations from missing at random conditional on treatment and baseline BPRS would be necessary to affect the conclusions.
* To address model misspecification, supplemental comparison of linear change in BPRS from baseline between treatment groups using the using Wilcoxon's rank-sum test and the Hodges-Lehmann estimate of location change with 95% confidence interval. In addition, model assumptions will be assessed by residual plots. Deviations from assumptions are not assumed to increase the Type I error, but may affect the interpretation of the estimated treatment contrast.
* To address non-adherence and protocol deviations, supplemental analysis using the primary model, for patients with two doses of treatment and no major protocol deviations up to 8 months, as determined at data base lock before unblinding.

BPRS at four months will be analyzed using the same method as for the primary time point, including sensitivity analyses. The main purpose of the four-month measurement is exploration of time to response.

SECONDARY EFFICACY OUTCOMES:

All analyses will be performed without formal multiplicity adjustment, for observed cases.

CGI-S over time will be presented by individual time series plots, and for each visit by number and percentage of patients in each category, and of patients satisfying the criteria for response (at least 2-point reduction from baseline), partial response (a 1 point reduction from baseline), and remission (CGI-S score 1-3). The categorical outcome response/partial response/no response will be analysed using logistic regression with randomized treatment as the only factor and presented as the common odds ratio with 95% CI and 2-sided p-value, at 8 months (primary time point) and at 4 months. Remission at the same time points will be analysed using logistic regression and presented as odds ratios with 95% CI and 2-sided p-value.

World Health Organization Disability Assessment Schedule (WHODAS) results will be presented as domain scores based on item response theory based scoring, and total disability score. Domain and total scores over time will be described using individual time series plots and mean value plots by randomized treatment. Domain and total scores, and linear change from baseline scores, at each time point will be described by randomized treatment using dot plots, scatter plots with baseline value on the x-axis, and tables of mean, standard deviation, median, min, max and quartiles. Total disability score at 8 months (primary) and 4 months will be analysed using a linear model with randomized treatment and baseline score as covariates and presented as mean difference with 95% CI and 2-sided p-value.

Yale Brown Obsessive Compulsion Scale (Y-BOCS) results will be presented and analyzed in the same way as WHODAS disability score. In addition, the number and proportion of patients with score 15 or below will be presented and analyzed in the same way as remission defined by CGI-S.

Bush-Francis Catatonia Rating Scale (BFCRS) total score over time will be described using individual time series plots and mean value plots by randomized treatment. Domain and total scores, and linear change from baseline scores, at each time point will be described by randomized treatment using dot plots, scatter plots with baseline value on the x-axis, and tables of mean, standard deviation, median, min, max and quartiles.

Pittsburgh Sleep Quality Index (PSQI) global sum will be tabulated descriptively by randomized treatment for each time point, using mean, standard deviation, median, quartiles, min and max, and number and percentage of patients with global sum 5 or higher.

EuroQol-5D (EQ-5D) domain scores will be presented for each time point using descriptive frequency tables and stacked bar charts by randomized treatment. EQ-5D Visual Analogue Scale (VAS) scale scores will be presented for each time point using descriptive tables of mean, standard deviation, median, min, max and quartiles.

Mismatch Negativity (MMN) amplitude and latency will be measured as the most negative data point within the 80-130 ms latency window, post-stimulus onset and compared between time points.

Biomarkers over time will be presented descriptively using individual time series plots and plots of geometric mean values over time by randomized treatment, and for each visit scatter plots with baseline on the x-axis and tables of geometric mean, geometric coefficient of variation (CV), median, quartiles, min and max, based on values over the limit of quantification, and number of observations under the limit of quantification. For infusion safety markers, the number and proportion of patients with values outside normal will also be tabulated. Biomarker concentrations at 8 months (primary) and 4 months will be analysed using a linear model for the log-transformed biomarker with randomized treatment and log-transformed baseline biomarker as covariates, and presented as the geometric mean ratio with 95% CI and two-sided p-value.

DETERMINATION OF SAMPLE SIZE Within- and between-patient standard deviation was estimated to 7.1 and 6.7 points respectively, from five case series with in total 35 measurements pre- and post-rituximab treatment, using a linear mixed-effect model with random intercept and rituximab treatment as a fixed factor.

Power was estimated using simulation. Baseline and 8 months BPRS were simulated with a 7 point standard deviation (SD) normally distributed random variation both within and between patients (corresponding to a total SD=9.8 points for a single measurement), and a homogenous treatment effect, using R v. 3.3.1. 40 patients, 20 patients per group, would give 81% power to detect an 8 point adjusted mean difference in BPRS between the rituximab and placebo groups, and 89% power to detect a difference of 9 points. Reasonable power would be retained under 5% random drop-out, with 79% power to detect an 8 point difference and 87% power to detect a 9 point difference between the groups. The power to detect a 9 point difference would still be 85% with 10% random drop-out.

ELIGIBILITY:
INCLUSION CRITERIA

General criteria

1. Diagnostic criteria: ICD 10 at least one of the following ICD 10 diagnoses:

   1. Obsessive-compulsive disorder ICD F42 or
   2. Obsessive-compulsive behavior ICD R46.81 AND/OR
   3. Schizophrenia, delusional, and other non-mood psychotic disorders, namely

   F20 Schizophrenia

   F22 Delusional disorders

   F23 Brief psychotic disorder

   F25 Schizoaffective disorders

   F28 Other psychotic disorder not due to a substance or known physiological condition

   F29 Unspecified psychosis not due to a substance or known physiological condition
2. Age: 18-55
3. Severity: Clinical Global impression (CGI): Minimum score of "4 = Moderately ill"
4. Swedish or English proficiency
5. The patient has tried at least 2 standard psychiatric medications at maximal tolerable or maximal recommended dosage for his/her current condition over a period of 6 months, but has not improved significantly
6. Medication has been unchanged for at least one month prior to study start
7. Signed informed consent
8. Use of adequate contraception
9. Radiological evidence of brain atrophy and scarring are absent
10. The clinical picture indicates active inflammatory activity (see specific criteria below), potential for rehabilitation and time from disease and/or episode debut is no longer than 10 years.

    Specific criteria
11. Acute (<12 weeks) or atypical debut, or episodes of any of the following:

    1. Symptoms of encephalopathy:

       psychotic symptoms, including hallucinations, delusions, paranoia, disorganized speech, disorganized behavior

       agitation, confusion

       sudden change in personality as perceived by the social environment

       drowsiness

       loss of functions in daily Life

       cognitive problems (memory, speech, learning)

       emotional dysregulation
    2. Focal neurological symptoms, e.g. ataxia, dystonia, myoclonus, sensory losses, paresthesia
    3. Psychomotor anomaly, e.g.retardation, catatonic symptoms, parkinsonism
    4. Loss of drive (sleep, appetite, libido, motivation)
    5. Obsessions, compulsions (OCD/OCB),
    6. Hypo- or hypervigilance (for e.g sounds, emotions, other peoples´ or own behavior)
    7. Sleeping disorders,

    AND
12. At least one of the following criteria:

    1. Prodromal phase with infection or symptoms of infection (fever, malaise, etc)
    2. Clinical improvement of psychiatric symptoms after treatment with anti-inflammatory medications other than antibody therapy (such as steroids, NSAIDs IVIG, plasmaphereses), or antibiotics
    3. Radiological evidence of neuroinflammation (MR)
    4. EEG pathology or witnessed epileptic seizure
    5. Biochemical evidence of inflammation, autoimmunity or blood-brain barrier dysfunction in blood or CSF samples, such as one of the following:

       presence of oligoclonal bands

       elevated CSF cell count

       elevated albumin quotient, or elevated albumin in CSF

       elevated Immunoglobulin G (IgG) ratio

       elevated levels of neurofilament
    6. Patient history of autoimmune disorder not associated with neuroinflammation, such as type 1 diabetes, rheumatoid arthritis, Sjögren´s syndrome, inflammatory bowel disease (IBD, comprising Crohn´s disease and ulcerative colitis), celiac disease, Grave´s disease, Hashimoto's thyroiditis
    7. Biochemical indication of autoimmunity such as elevated serum anti-thyroid peroxidase (TPO) antibody, antinuclear antibody (ANA), anti-neutrophil cytoplasmic antibody (ANCA), rheumatoid factor (RF) or glutamic acid decarboxylase (GAD) antibodies, PANDAS panel with relationship to symptom development.

    EXCLUSION CRITERIA
13. Concomitant malignancies or previous malignancies within the last five years
14. Cannot comply with vaccination recommendations
15. History of severe allergic or anaphylactic reactions in conjunction with prior treatment with monoclonal antibodies
16. Prior antibody therapy including Rituximab (MabThera®/Rituxan®)
17. Patient has been treated with clozapine (which may have immunosuppressant effect), systemic corticosteroids or IVIG within 60 days prior to screening visit
18. Prior treatment with immunosuppressant medications (not including systemic corticosteroids and IVIG) for other medical condition
19. History of or positive screening for HIV, Tuberculosis, Hepatitis B and/or Hepatitis C (ever)
20. Heart disease such as previous heart attack, arrhythmia or heart failure, coronary insufficiency
21. Current drug, alcohol, or chemical abuse
22. Pregnancy at any time during the study
23. Known chronical significant bacterial/viral/fungal infections at infusion date
24. Diagnosis of well-established neuroinflammatory disease such as Multiple Sclerosis (MS) (ICD codes G00-G09, G35-G37) or systemic lupus erythematosus (SLE) (M32)
25. Tested positive for autoantibodies in serum or CSF associated to known and treatable neuroinflammatory disease (such as neuroborreliosis, treatable autoimmune encephalitis). Patients having completed recommended treatment without significant improvement may still be included in this study.
26. History of any illness that in the opinion of the investigator may jeopardize the ability of the patient to participate in the study.
27. Patient is enrolled in another medical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
BPRS | 8 months
  Brief Psychiatric Rating Scale, is a broad psychiatric interview and evaluation tool comprising 24 items, of which 14 are rated based on the individual´s self-report, and ten based on observed behavior and speech. Each item is rated 1 to 7 (1 = not present, 7 = extremely severe). Minimum score with all items assessed is 24, maximum score is 168. Higher score signifies higher degree of psychiatric symptoms i.e. worse outcome. Primary outcome measure is the mean difference in total score between the trial arms at 8 months.

SECONDARY OUTCOMES:
WHODAS | baseline, 4 months, 8 months, 12 months, 16 months
  World Heath Organization Disability Assessment Schedule (36 questions self-rated by participant). Each item is assigned a score from 1 ("none") to five ("extreme"). Minimum score is 36, maximum score 180 with higher score meaning worse outcome.
CGI | baseline, 4 months, 8 months, 12 months, 16 months
  Clinical global impressions of severity (CGI-S) and improvement (CGI-I) as rated by investigator. Severity of illness (CGI-S) is rated from 1 = "normal, not ill" to 7 = "among the most extremely ill patients", i.e. higher score means worse outcome. Global improvement (CGI-I) is rated from 1 = "Very much improved" to 7 = "Very much worse" i.e. higher score meaning worse outcome.
EQ-VAS | baseline, 4 months, 8 months, 12 months, 16 months
  EuroQol Visual analogue scale; measures self-rated health on a visual analogue scale. Score ranges from 0 to 100, with higher score meaning better outcome.
Y-BOCS | baseline, 4 months, 8 months, 12 months, 16 months
  Yale Brown Obsessive Compulsive Scale; using 10-item investigator-administered assessment of the frequency of obsessions and compulsions. Each item is scored from 0 to 4, with higher score indicating more severe symptoms i.e. worse outcome. Minimum score is 0, maximum is 40.
BFCRS | baseline, 4 months, 8 months, 12 months, 16 months
  Bush Francis Catatonia Rating Scale, an investigator-rated 23-item scale for catatonic signs and their severity. Each item is rated from 0 to 3 (items 13, 17, 18, 19, 20 and 21 can only be assigned 0 or 3), with higher score indicating more severe symptoms, i.e. worse outcome. Minimum score is 0, maximum is 69.
MMN | baseline, 8 months, 16 months
  Mismatch negativity (MMN); measuring differences in brain reactions to infrequently ("deviant") vs frequently occuring ("standard") auditory stimuli. EEG is recorded during a 12-minute session with the patient listening to an odd-ball paradigm of 1440 standard tones and 360 duration variants. 400 ms-windows are averaged and the maximum difference in negativity between standards and deviants is recorded as the MMN.
  MMN amplitude and latency will be measured as the most negative data point within the 80-130 ms latency window, post-stimulus onset and compared between time points. Previous data is not available for this population.
Neurological exam | baseline, 8 months, 16 months
  The following items will be examined and judged normal or abnormal. Outcome is change in number of pathological items over time. More abnormal items means worse outcome.
  * dysarthria
  * dysphasia
  * verbal coherence
  * awareness of person, place and time
  * involuntary movements
  * walking pattern
  * heel-to-toe gait
  * heel walking and toe walking
  * squatting and raising up
  * knee extension
  * tone of knee joints, elbows, wrists
  * reflexes: patellar, achilles, biceps, triceps
  * plantar response (Babinski´s sign)
  * heel-to-shin-test
  * finger-to-nose test
  * diadochokinesis
  * light-touch sensation on hands and feet
  * pin-prick sensation on hands and feet
  * vibration sensation on ankles and wrists
  * eye movement (including nystagmus, ptosis)
  * pupil size and reaction to light
  * Donder´s field-of-view-test
  * friction sound hearing test
  * facial motor functions
  * uvula asymmetry
  * tongue motor functions
  * finger and shoulder abduction
  * Grassets test
  * Rombergs test
Change in plasma/serum and CSF markers for immune activity | baseline, 8 months, 16 months
  The concentration of diverse markers for immune activity e.g. autoantibodies, cytokines, chemokines, immunoregulatory molecules, will be measured at baseline, 8 months and 16 months.
  Biomarker concentrations over time will be presented descriptively using individual time series plots, and plots of geometric mean values over time by randomized treatment. The exact biomarkers to be analyzed will be specified before data collection for this study is completed and before the code is broken.
BPRS | 4 months, 12 months, 16 months
  Brief Psychiatric Rating Scale, is a broad psychiatric interview and evaluation tool comprising 24 items, of which 14 are rated based on the individual´s self-report, and ten based on observed behavior and speech. Each item is rated 1 to 7 (0 = not assessed, 1 = not present, 7 = extremely severe). Minimum score with all items assessed is 24, maximum score is 168. Higher score signifies higher degree of psychiatric symptoms i.e. worse outcome. BPRS at 4, 12 and 16 months will be analyzed using the same method as for the primary time point.
SWM | baseline, 8 months, 16 months
  CANTAB digital version of Spatial Working Memory (SWM). Among a number of digital colored squares, participants are to find yellow tokes and use them to fill up an empty column. Outcome is measured by number of errors (revisiting squares), with higher error number meaning worse outcome.
RTI | baseline, 8 months, 16 months
  CANTAB digital version of Reaction Time (RTI). Participants must react as soon as possible to indicate a yellow dot that appears in one of five circles. Outcome measures are divided into reaction time and movement time. Longer time means worse outcome.
PAL | baseline, 8 months, 16 months
  CANTAB digital version of paired associates learning (PAL). Several boxes displayed on a screen. Some of them contain a pattern. Participants must allocate a displayed pattern to the correct box. Outcome is measured by number of errors (higher number means worse outcome), number of trials required to locate pattern(s) correctly (higher number means worse outcome), memory scores (higher score means better outcome) and stages completed (more stages means better outcome).
MTT | baseline, 8 months, 16 months
  CANTAB digital version of Multitasking Test (MTT). The test displays an arrow which can appear on either the right or left side of the screen, and can point either to the right or to the left.
  A cue at the top of the screen indicates to the participant which rule they are to follow to select the right or left button: either according to "the side on which the arrow appeared" or according to "the direction in which the arrow was pointing".
  Outcome measures include response latencies and error scores. Longer latency and higher error score mean worse outcome.
OTS | baseline, 8 months, 16 months
  CANTAB digital version of One Touch Stockings of Cambridge (OTS). The participant is shown an upper and a lower display containing three colored balls each. The participant is to work out in their head how many moves that are required to copy the pattern in the upper display to the lower display. Outcome measures are number of problems solved on first choice (higher number means better outcome), mean choices to correct (higher number means worse outcome), speed of response to first choice (if the first choice was correct, longer time means worse outcome) and mean latency to correct (loger latency means worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Janet L Cunningham, MD PhD, Principal Investigator — Uppsala University Hospital and Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Debnath M, Venkatasubramanian G. Recent advances in psychoneuroimmunology relevant to schizophrenia therapeutics. Curr Opin Psychiatry. 2013 Sep;26(5):433-9. doi: 10.1097/YCO.0b013e328363b4da. PMID 23867655
- [Background] Attwells S, Setiawan E, Wilson AA, Rusjan PM, Mizrahi R, Miler L, Xu C, Richter MA, Kahn A, Kish SJ, Houle S, Ravindran L, Meyer JH. Inflammation in the Neurocircuitry of Obsessive-Compulsive Disorder. JAMA Psychiatry. 2017 Aug 1;74(8):833-840. doi: 10.1001/jamapsychiatry.2017.1567. PMID 28636705
- [Background] Brimberg L, Benhar I, Mascaro-Blanco A, Alvarez K, Lotan D, Winter C, Klein J, Moses AE, Somnier FE, Leckman JF, Swedo SE, Cunningham MW, Joel D. Behavioral, pharmacological, and immunological abnormalities after streptococcal exposure: a novel rat model of Sydenham chorea and related neuropsychiatric disorders. Neuropsychopharmacology. 2012 Aug;37(9):2076-87. doi: 10.1038/npp.2012.56. Epub 2012 Apr 25. PMID 22534626
- [Background] Lee WJ, Lee ST, Byun JI, Sunwoo JS, Kim TJ, Lim JA, Moon J, Lee HS, Shin YW, Lee KJ, Kim S, Jung KH, Jung KY, Chu K, Lee SK. Rituximab treatment for autoimmune limbic encephalitis in an institutional cohort. Neurology. 2016 May 3;86(18):1683-91. doi: 10.1212/WNL.0000000000002635. Epub 2016 Apr 1. PMID 27037228
- [Background] Dazzi F, Shafer A, Lauriola M. Meta-analysis of the Brief Psychiatric Rating Scale - Expanded (BPRS-E) structure and arguments for a new version. J Psychiatr Res. 2016 Oct;81:140-51. doi: 10.1016/j.jpsychires.2016.07.001. Epub 2016 Jul 4. PMID 27451107